CLINICAL TRIAL: NCT06209177
Title: A Phase 1/2a Dose-Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ARO-CFB in Adult Healthy Volunteers and Adult Patients With Complement-Mediated Kidney Disease
Brief Title: Study of ARO-CFB in Adult Healthy Volunteers and Patients With Complement-Mediated Kidney Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROCFB-1001
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1, participants are randomized to receive either ARO-CFB or placebo. Participants, care providers, investigator and outcomes assessors are all blinded to treatment assignment. Part 2 in patients with IgAN is open-label and there is no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ARO-CFB (Healthy Volunteers) (Experimental): 1 or 2 doses of ARO-CFB by subcutaneous (sc) injection
  Interventions: Drug: ARO-CFB
- Placebo (Healthy Volunteers) (Experimental): placebo calculated volume to match active treatment by sc injection
  Interventions: Drug: Placebo
- ARO-CFB (Adult Patients with IgAN) (Experimental): 3 doses of ARO-CFB by sc injection
  Interventions: Drug: ARO-CFB

INTERVENTIONS:
Drug: ARO-CFB — ARO-CFB for sc injection
  Arms: ARO-CFB (Adult Patients with IgAN); ARO-CFB (Healthy Volunteers)
Drug: Placebo — sterile normal saline (0.9% NaCl for sc injection)
  Arms: Placebo (Healthy Volunteers)

SUMMARY:
The purpose of AROCFB-1001 is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ARO-CFB Injection in adult healthy volunteers (HVs) and in adult patients with complement-mediated kidney disease (IgA Nephropathy [IgAN]). In Part 1 of the study, HVs will receive either one or two doses of ARO-CFB or placebo. In Part 2 of the study, adult patients with IgAN will receive 3 open-label doses of ARO-CFB. Dose levels in Part 2 will be determined based on cumulative safety and pharmacodynamic data from Part 1.

ELIGIBILITY:
Inclusion Criteria (All Participants):

* Willing to provide written informed consent and to comply with study requirements
* Female participants must be non-pregnant/non-lactating
* Healthy volunteers must be willing to be vaccinated with a meningococcal and pneumococcal vaccine. IgAN participants must have been vaccinated or willing to undergo vaccination
* All participants must be willing to be vaccinated or have a history of vaccination for Haemophilus influenzae type B
* Body Mass Index (BMI) between 18.0 and 35.0 kg/m2
* Participants of childbearing potential must agree to use highly effective contraception in addition to a condom during the study and for at least 90 days following the end of the study or the last dose of study drug, whichever is later. Participants must not donate sperm or eggs during the study and for at least 90 days following the end of the study or last dose of study drug, whichever is later.
* No abnormal finding of clinical relevance at the Screening evaluation that, in the opinion of the Investigator, could adversely impact participant safety or adversely impact study results.

Inclusion Criteria (IgAN Participants):

* Diagnosis of IgA Nephropathy based on renal biopsy within 5 years
* Clinical evidence of ongoing disease based on significant proteinuria
* Estimated glomerular filtration rate ≥30 mL/min/1.73m2 at Screening and currently not on dialysis
* Must have stable or worsening renal disease, on stable and optimized treatment for at least 30 days prior to Screening and willing to stay on a stable standard of care regimen for the duration of the study
* Must be on a maximally recommended or tolerated dose of an angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB)

Exclusion Criteria (All Cohorts):

* History of recurrent or chronic infections including infections caused by encapsulated bacterial organisms or viruses
* History of active bacterial, viral, or fungal infection within 14 days prior to treatment administrations
* Seropositive for Human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
* History of meningococcal infection
* History of asplenia
* History of severe aplastic anemia or concurrent severe aplastic anemia
* Known or suspected hereditary complement deficiency or other primary immunodeficiency syndrome
* History of diabetes mellitus (Type 1 or Type 2)
* Uncontrolled hypertension

Exclusion Criteria (IgAN Participants):

* Nephrotic syndrome or rapidly progressive glomerulonephritis
* Suspicion for secondary etiologies of IgAN
* Evidence of non-IgAN kidney disease on renal biopsy
* Renal biopsy showing interstitial fibrosis/tubular atrophy of more than 50%
* Use of complement inhibitors or monoclonal antibody therapies for treatment of IgAN

Note: Additional Inclusion/Exclusion criteria may apply per protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (AEs) and/or Serious Adverse Events (SAEs) | Part 1: up to Day 169 (End of Study [EOS]); Part 2: up to Day 225 (EOS)

SECONDARY OUTCOMES:
Change from Baseline in Serum Complement Factor B (CFB) and Its Breakdown Products Ba and Bb | Part 1: up to Day 169 (End of Study [EOS]); Part 2: up to Day 225 (EOS)
Pharmacokinetics (PK) of ARO-CFB: Maximum Observed Plasma Concentration (Cmax) | Part 1 only: up to 48 hours postdose
PK of ARO-CFB: Time to Maximum Observed Plasma Concentration (Tmax) | Part 1 only: up to 48 hours post-dose
PK of ARO-CFB: Area Under the Plasma Concentration Versus Time Curve from Zero to 24 Hours (AUC0-24) | Part 1 only: up to 48 hours post-dose
PK of ARO-CFB: Area Under the Plasma Concentration Versus Time Curve from Zero to the Last Quantifiable Plasma Concentration (AUClast) | Part 1 only: up to 48 hours post-dose
PK of ARO-CFB: Area Under the Plasma Concentration Versus Time Curve from Zero Extrapolated to Infinity (AUCinf) | Part 1 only: up to 48 hours post-dose
PK of ARO-CFB: Terminal Elimination Half-Life (t1/2) | Part 1 only: up to 48 hours post-dose
PK of ARO-CFB: Apparent Clearance (CL/F) | Part 1 only: up to 48 hours post-dose
PK of ARO-CFB: Volume of Distribution (Vz/F) | Part 1 only: up to 48 hours post-dose
PK of ARO-CFB: Amount of Drug Recovered in Urine Over Zero - 24 Hours Post-dose (Ae) | Part 1 only: up to 24 hours post-dose
PK of ARO-CFB: Fraction of Drug Excreted Unchanged (fe) | Part 1 only: up to 24 hours post-dose
PK of ARO-CFB: Renal Clearance (CLr) | Part 1 only: up to 24 hours post-dose
Percent Change from Baseline in Serum Complement Factor B (CFB) and Its Breakdown Products Ba and Bb | Part 1: up to Day 169 (End of Study [EOS]); Part 2: up to Day 225 (EOS)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No